CLINICAL TRIAL: NCT01631396
Title: Comparison of Two Neuromuscular Anesthetics Reversal in Obese Patient Undergoing Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Sponsor
Other Study IDs: AR-002-12
Record Dates: First submitted 2012-06-14; First posted 2012-06-29 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2012-03

CONDITIONS: Anesthesia; Surgery
Keywords: Morbid obesity; Bariatric Surgery; Neuromuscular block reversal
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients recieving Sugammadex: Sugammadex Group (n=20) - anesthesia induced by Rocuronium 0.4mg/kg body, additional Rocuronium 0.1-0.2 mg/kg body as needed during surgery (not more than x2), muscular blockage reversal using Sugammadex 2.0 mg/kg body.
  Interventions: Drug: Sugammadex vs. Neostigmine
- Patients recieving Neostigmine: Neostigmine Group (n=20) - anesthesia induced by Rocuronium 0.4mg/kg body, additional Rocuronium 0.1-0.2 mg/kg body as needed during surgery (not more than x2), muscular blockage reversal using Neostigmine 0.05 mg/kg body and atropine 0.1 mg/kg body.
  Interventions: Drug: Sugammadex vs. Neostigmine

INTERVENTIONS:
Drug: Sugammadex vs. Neostigmine — * Sugammadex Group (n=20) - anesthesia induced by Rocuronium 0.4mg/kg body, additional Rocuronium 0.1-0.2 mg/kg body as needed during surgery (not more than x2), muscular blockage reversal using Sugammadex 2.0 mg/kg body.
  * Neostigmine Group (n=20) - anesthesia induced by Rocuronium 0.4mg/kg body, additional Rocuronium 0.1-0.2 mg/kg body as needed during surgery (not more than x2), muscular blockage reversal using Neostigmine 0.05 mg/kg body and atropine 0.1 mg/kg body.

SUMMARY:
The study is a prospective, single center, double arm study aiming at the comparison of 2 commercial neuromuscular block reversal drugs: Neostigmine (Cooper S.A.) and Sugammadex (MSD). A faster recovery from neuromuscular block is expected for patients receiving Sugammadex and this protocol is of high importance for anesthesia of morbid obese patients during bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Morbidly obese male or female patients in the age 20-65 that are candidates for bariatric surgery.
2. Patients that can read and understand the fundamental nature of the clinical protocol.
3. Patients must sign the Informed Consent Form.

Exclusion Criteria:

1. Patients treated with drugs that might interact with Rocuronium.
2. Patients with history of malignant hyperthermia.
3. Patients with significant renal disease.
4. Patients with a known allergy to one of the drugs used during anesthesia.
5. Patients with known muscular disease.
6. Patients with severe cardiovascular disease (NYHA>2)
7. Breast feeding patients
8. Patients refusing to follow the clinical protocol.
9. Patients participating in a different clinical trial.
10. Patients refusing to sign the Informed Consent Form
11. Physician's objection.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects for the study will be recruited from patients within the community who have sought treatment for morbid obesity by bariatric surgery, are qualified for the surgery and meet all of the eligibility criteria listed below.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Safety of Sugammadex reversal - number of drug-related adverse events with Sugammadex <= that of Neostigmine. | Monitoring nueromuscular reaction from end of anesthesia recovery (in the OR) intil patient is released from hospital (48-72 h post surgery)
  The number of drug-related adverse events using Sugammadex is smaller or equal to those using Neostigmine.

SECONDARY OUTCOMES:
Use of Sugammadex for neuromuscular anaesthesia reversal higher patient satisfaction compared to Neostigmine. | Monitoring nueromuscular reaction from end of anesthesia recovery (in the OR) intil patient is released from hospital (48-72 h post surgery)
  Neuromuscular anesthesia reversal with Sugammdex is fast, comfortable and well accepted by the patients. Time of recovery from anesthesia and patient satisfaction will be compared for the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Asnat Raziel, MD, Principal Investigator — Medical Director, ICBS-Israeli Center for Bariatric Surgery
Locations (1):
- Assuta Medical Center, Tel Aviv, Israel